CLINICAL TRIAL: NCT00829595
Title: Pneumococcal Vaccination in Patients With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Gil Melmed, MD, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6355
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Inflammatory Bowel Disease; Crohn Disease; Ulcerative Colitis
Keywords: inflammatory bowel disease; Crohn disease; ulcerative colitis; immunosuppression; anti tumor necrosis alpha; pneumovax; pneumococcal vaccine
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): IBD, on both an anti-TNF agent and an immunomodulator
  Interventions: Biological: 23-valent polysaccharide pneumococcal vaccine (Pneumovax TM)
- 2 (Experimental): IBD, not on any immunosuppressive medications
  Interventions: Biological: 23-valent polysaccharide pneumococcal vaccine (Pneumovax TM)
- 3 (Active Comparator): Healthy, non-IBD, not on immunosuppressive medications (control arm)
  Interventions: Biological: 23-valent polysaccharide pneumococcal vaccine (Pneumovax TM)

INTERVENTIONS:
Biological: 23-valent polysaccharide pneumococcal vaccine (Pneumovax TM) — 0.5mL intramuscular, one time
  Other Names: Pneumovax

SUMMARY:
Patients with inflammatory bowel disease (IBD) will be assessed for immunologic response to pneumococcal vaccination. Patients with IBD meet criteria as outlined by the Centers for Disease Control (CDC) for pneumococcal vaccination, yet the investigators have found that pneumococcal vaccination in this population is under-utilized. It is unknown whether or not IBD or IBD-related medications impact the immune response to this recommended vaccine.

Three groups of 25 patients each will be recruited. The first group will consist of outpatients with IBD who are receiving infliximab (Remicade TM) while on concommitant immunosuppressive therapy (with either 6MP, azathioprine, or methotrexate). This group is intended to represent a common 'heavily immunosuppressed' patient group with IBD.

The second group will consist of patients with IBD seen in our outpatient clinic who are not on any immune-suppressive medications. These patients meet CDC criteria for vaccination by virtue of having a chronic medical illness. The third group will consist of healthy age-matched (to the first group) controls.

After obtaining informed consent, patients will be screened with baseline lab tests including testing for antibodies against pneumococcus. At the baseline visit, patients will also undergo a brief medical history, physical examination, and assessment of their IBD disease activity.

Included patients will then undergo a one-time intramuscular vaccination with 23-valent polysaccharide pneumococcal vaccine (Pneumovax TM). One month later, subjects will return for a blood draw to assess for response to pneumococcal vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females over the age of 18 with inflammatory bowel disease; healthy controls will be age- and sex-matched.
2. The patient must understand and voluntarily sign and informed consent document
3. A history of chronic (greater than 1 month) ulcerative colitis or Crohn's disease diagnosed and documented by the standard clinical, radiographic, endoscopic, and histopathologic criteria
4. (Group 1): Outpatients at CSMC IBD center with IBD who are on maintenance anti-TNF therapy with infliximab OR ADALIMUMAB plus concomitant immunomodulator therapy (with either 6MP, AZA, or MTX)
5. (Group 2): Outpatients at CSMC's IBD Center with documented IBD who are not on any immune-suppressive medications. Treatment with oral or topical 5-ASA products, antibiotics, or probiotics, are permitted.
6. (Group 3): Healthy volunteers without chronic illness, not on immune-suppressive medications.

Exclusion Criteria:

1. Hypersensitivity to any component of the vaccine
2. Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, endocrine (including thyroid), pulmonary, cardiac, infectious, neurologic or cerebral disease. Included are ongoing chronic active conditions such as chronic active hepatitis.
3. Patients who in the judgment of the investigator are unwilling or unable to comply with all the protocol-related assessments and procedures.
4. History of alcohol or other drug abuse within one year, or any conditions associated with poor compliance.
5. Patients in whom venipunctures are not feasible due to poor tolerability or lack of easy access.
6. Healthy volunteers or patients with a history of prior pneumococcal vaccination
7. Any condition which, in the opinion of the Investigator, places the patient at unacceptable risk if he/she were to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Response, defined by postvaccination antibody titers | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Vasiliauskas, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States